CLINICAL TRIAL: NCT00873691
Title: Prospective Comparison of 50/50% Tilt and Tuned Defibrillation Waveforms in Right-Sided Implants
Brief Title: Comparison of Fixed Tilt and Tuned Waveforms in Right-sided Implants
Acronym: Tilt & Tune
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD 442
Record Dates: First submitted 2009-03-30; First posted 2009-04-01 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Patients indicated for an ICD/ CRT-D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: ICD shocks programmed to Tuned Waveform
  Interventions: Device: ICD
- 2: ICD shocks programmed to 50% Tilt waveform
  Interventions: Device: ICD

INTERVENTIONS:
Device: ICD — Intervention isn an ICD. Patients in experimental group will have their ICDs programmed to Tuned waveform and those in the control group will have their ICDs programmed to Fixed Tilt waveform.

SUMMARY:
The purpose of this study is to compare the defibrillation efficacy between the 50/50% tilt biphasic waveform and the Tuned biphasic waveform in patients with right-sided implants.

DETAILED DESCRIPTION:
Current era implantable cardioverter defibrillators (ICDs) have high defibrillation efficacy. This has stimulated a debate about whether DFT testing should be performed at all.1-3 However, this dialog has primarily centered around left sided implants, a group that is characterized by a small incidence of high defibrillation thresholds (DFTs).

The mechanism of phase duration programming to improve DFTs would seem to be most effectively applied to a group of patients with a high incidence of high DFTs such as right sided implants. This study therefore aims to prospectively evaluate direct phase duration programming on DFTs in right sided implants.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets standard indication for an ICD/ CRT-D
* Patient will be implanted with an FDA approved SJM ICD/ CRT-D that has a higher capacitance (maximum delivered energy - 36 J)
* Pulse generator will be implanted on the right-side
* Patient is able to tolerate DFT testing.
* RV lead will be placed in the RV apex or inferior septum

Exclusion Criteria:

* Patient is pregnant.
* Patient is less than 18 years old.
* SVC coil was turned ON during DFT testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with approved ICD/CRT-D indications
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2009-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
True Design for Test (DFTs) in fixed tilt and tuned waveforms obtained in volts (V) | Baseline

SECONDARY OUTCOMES:
True DFTs in fixed tilt and tuned waveforms obtained in joules (J) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Varma, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Varma N, Efimov I. Right pectoral implantable cardioverter defibrillators: role of the proximal (SVC) coil. Pacing Clin Electrophysiol. 2008 Aug;31(8):1025-35. doi: 10.1111/j.1540-8159.2008.01130.x. PMID 18684259
- [Background] Natarajan S, Henthorn R, Burroughs J, Esberg D, Zweibel S, Ross T, Kroll M, Gianola D, Oza A. "Tuned" defibrillation waveforms outperform 50/50% tilt defibrillation waveforms: a randomized multi-center study. Pacing Clin Electrophysiol. 2007 Jan;30 Suppl 1:S139-42. doi: 10.1111/j.1540-8159.2007.00624.x. PMID 17302691
- [Derived] Varma N, Schaerf R, Kalbfleisch S, Pimentel R, Kroll MW, Oza A. Defibrillation thresholds with right pectoral implantable cardioverter defibrillators and impact of waveform tuning (the Tilt and Tune trial). Europace. 2017 Nov 1;19(11):1810-1817. doi: 10.1093/europace/euw306. PMID 27986795